CLINICAL TRIAL: NCT02489877
Title: Comparison Between Clinical and MRI Multiple Sclerosis Activity and Expression of Human Endogenous Retrovirus Type W and Herpesvirus in Peripheral Blood of Patients
Brief Title: Comparison Between Clinical and MRI Multiple Sclerosis Activity and Expression of Human Endogenous Retrovirus Type W and Herpesvirus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Guilherme Sciascia do Olival, expert - medical residence, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: Fcmscsp-HERV
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; HERV-W virus; Herpesviridae family
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Multiple Sclerosis: Patients diagnosed with Multiple Sclerosis
- without Multiple Sclerosis: Healthy individuals without neurological disease associated
- with other neurological diseases: Patients diagnosed with the following diseases: Lateral Amniotrofic Sclerosis, Headache , Parkinson's disease, Dementia and Epilepsy.

SUMMARY:
Multiple sclerosis is the most common autoimmune inflammatory disease of the central nervous system. It is known that your etiology has genetic and environmental causes. Several viruses have been implicated as triggers as well as perpetrators of this disease. Several studies make the correlation between Endogenous Retrovirus Type W (HERV-W) and the family Herpesviridae and activity in the pathogenesis of multiple sclerosis. The most important characteristics of the virus implicated in the pathogenesis of the disease is the fact that they have latency periods of exacerbation and they have, as their main biological environment, the central nervous system. The HERV-W, Epstein-Barr virus (EBV), cytomegalovirus, herpes virus type 6 and type 7 herpesvirus members are the most studied as causes of multiple sclerosis. It was found that these viruses are closely involved in the pathogenesis of MS, but it is believed that aren't the only responsible for its beginning. It is likely that this disease presents numerous triggers and more studies are needed to determine these interactions. In addition, a study comparing the activity of multiple sclerosis with the presence of these viruses was never realized.

DETAILED DESCRIPTION:
Background/Rationale:

Multiple Sclerosis (MS) is an inflammatory demyelinating disease that affects the spinal cord (especially in posterior cords). The clinical heterogeneity of MS is well described, but currently it is known that lesions of MS and mechanisms underlying involved in the pathological destruction of the central nervous system (CNS) are also heterogeneous. It is a multifactorial disease in which one immunopathogenic mechanism is suggested as responsible for the destruction of the sheath myelin.

However, the pathology of inflammatory joint lesions of MS suggests that specific autoimmune responses against components of CNS myelin may have a crucial role in the destruction of myelin. This concept is supported by the high level of oligoclonal immunoglobulin G (IgG) in cerebrospinal fluid by linkage with the locus of the major histocompatibility complex (MHC), expansion of B and T cells reactive to myelin in MS lesions and the fact that immunization with myelin proteins induces an MS-like disease in animals, experimental autoimmune encephalomyelitis (EAE).

The autoreactivity for various myelin proteins, including myelin basic protein, proteolipid protein, and myelin-associated glycoprotein in myelin oligodendrocyte glycoprotein (MOG), has been observed in patients with MS.

It is noted however, that T cells of patients with MS show a predominant activity against MOG in relation to other myelin proteins, and anti-MOG antibodies were identified connected to the myelin's disintegration around axons in acute lesions of MS. In addition, sensitization with MOG reproduces the clinical and demyelinating degenerative pathology of MS in rodent models and primates.

An infectious etiology of MS has also been postulated, and over several years, a number of different viruses have been suggested to trigger immunopathology. Increased titles of antibody were detected, for EBV, varicella zoster virus and rubella virus, while specific proteins human endogenous retroviruses (HERV), in particular of the HERV-W family were detected in the blood and brain lesions in patients with MS.

HERV arose from ancient infections of host cells of the germline by exogenous retroviruses and today constitute about 8% of the human genome.

The retrovirus multiple sclerosis-associated (MRSV), is an enveloped virus with reverse transcriptase activity, which represents the prototype of the HERV-W family human genome.

The MRSV was isolated in leptomeninges, in choroid plexus and in cultures of monocytes/macrophages of MS patients and their origin is still under investigation. Has been suggested that particles are originated from MSRV provirus HERV-W modified, or transmitted from a member of the same exogenous family. MSRV virions has properties such as superantigens, they induce the production of cytokines by mononuclear cells in peripheral human blood.

HERV particles associated with reverse transcriptase activity (RT) were confirmed to be a hallmark of expression from MSRV. A protocol for detection of MSRV virion by RT PCR was designed to detect their presence in serum and cerebrospinal fluid (CSF) of the patient .

Independent studies in patients with MS and control populations showed correlations between the MS and MSRV and its prognosis, including the conversion of relapsing-remitting MS in its secondary progressive form (SP-MS).

Parallel studies showed the immunopathogenesis of MSRV virions and identified the envelope protein (Env) of MSRV as being responsible for the pro-inflammatory and superantigenicity immune. The Env antigen was detected on MS patients in studies of brain postmortem.

The trans-activation of the HERV-W promoters by environmental virus associated with MS has also been shown to induce an epigenetic dysregulation in HERV-W, when present in the host genome.

Certainly the most important herpes virus associated with MS is EBV, the ratio between EBV serology and the development of MS has been extensively studied. Furthermore, the interaction between EBV and the immune system are undeniable leading to a persistent immune response and immortalization of lymphocytes. There are also studies that correlate the expression of EBV with greater activity of MS. Finally, the interaction between EBV and endogenous retroviruses are a recent and fascinating field of study.

EBV was the first member of the Herpesviridae family to be implicated as a potential cause of MS in 1971. EBV is a possible candidate due to several factors: it is widespread in nature, requires a long quiescent viral infection that has continuous production due periods of reactivation and modulate the human immune system.

The difficulty in associating MS to prove that EBV is the virus infection occurred before the onset of autoimmune disease. Pohl et al. showed that the EBV-seropositivity in patients with MS in Europe (children) - was 99% higher when compared with the control group, which virus antibodies were found in 72%.

Levin et al. estimated the time of viral infection by serum antibody titers before the MS and compared with a control group. This study had access to the medical records of approximately 8 million employees of the US Army who had stored blood samples. Of this group, the case-control study where 305 people came to later develop MS and 610 control subjects selected were paired; 10 cases who developed MS and 32 controls were initially EBV seronegative. All cases had become positive EBV before the MS, compared to only 35.7% of controls who seroconverted.

Other studies have also attempted to assess the relationship between antibody titers against EBV and the onset of MS. According to the work of De Lorenze et al., patients with MS had a significant increase in antibodies 20 years before the first symptoms of MS. This fact can be explained in two ways: the existence of a prior infection altering the balance of the EBV receptor cells (memory T cells) or reinfection with a different strain of EBV.

EBV infects B lymphocytes and persistently highly immunogenic. The antigen specific cytotoxic T lymphocytes are produced continuously and increased in number in response to primary infection and high viremia. This immune control is essential to prevent EBV-related malignancies. In its modulating action, manages to rescue infected B lymphocytes via expression of latent antigens and helps them to differentiate into memory B cells, where the virus persists. However, it is not established whether the increased T cells specific for EBV is a response to increased stimulation by specific recognition of myelin antigens. EBV viral load is not very high in MS, in addition, T cells specific for this virus does not seem to be distinguished from the same cells in hosts without MS.

Another investigator states that during periods of MS reactivation there is an increased activity of virus replication in relation to periods of remission. Patients with antibody response to early antigen of EBV are more likely to show disease activity as measured by MRI with gadolinium, when compared to patients without humoral response. These data led us to believe that the activity of the disease may be related to latent EBV infection as well as disease progression.

Studies correlating levels of antibodies against cytomegalovirus (CMV) and MS are controversial. Although most of the results show high rates of CMV infection in patients with MS, on the other hand, a milder presentation of the disease is observed.

Some investigators looked for the presence of anti-CMV antibodies in MS and healthy individuals. They found positive in 98% of MS patients compared with 52% in the control group.

Another investigators showed that patients who had antibody against CMV were: later age of disease onset, lower rates of reactivation of the disease, and fewer signs of cerebral atrophy on MRI. Those who had higher titers of these antibodies had less brain atrophy and fewer lesions on imaging tests, compared with patients who had lower titers. An animal model with mimic the patterns of MS demonstrated that animals with CMV infections demyelinating frame before clinical presentations were weaker than those not infected. These studies suggest a beneficial modulating effect of CMV infection on the immune response in MS.

The herpesvirus (HHV-6 and HHV-7) are closely related and have a similar biological pattern. These viruses are able to infect cells of the immune system and modulate their functions. The work described by Krukle-Nora et al. attempted to investigate associations between HHV-6 and HHV-7 in MS by analyzing the peripheral blood of patients. Patients were randomly selected and divided into 02 groups: 14 patients with relapsing remitting MS (RR-MS) and 14 with secondary progressive MS (SP-MS). All study patients were at least 3 months without use of immunosuppressive drugs. Of the 28 patients, 25 had latent HHV-6 infection and/or HHV-7. HHV-6 has been found in 9 patients with RR-MS and 9 with the SP-MS. HHV-7 were found in 10 patients with RR-MS and 14 with the SP-MS.

Two investigators using the technique of fluorescent in situ hybridization, human cadaveric tissues examined to evaluate the expression of early and late viral genes at white matter in the affected tissue of patients with MS and in brain samples without disease. The gene of HHV-6 was found in all samples and was restricted to oligodendrocytes. Quantitative analysis of the expression of viral RNA showed that in both groups of MS patients (brain tissue with and without change of white matter) samples had significantly higher levels of expression of this virus. Furthermore, they showed that the injured tissues were correlated with higher viral expression, a fact that contributes to the theory of HHV-6 is implicated in the pathogenesis of MS.

Using all these methods for virus were observed conflicting results. In fact when the technologies used were not capable of distinguishing active from latent infection by HHV-6 (by analysis of leukocytes from the blood, of cerebrospinal fluid containing cells and of tissue of the CNS), no difference is found among the samples patients and the control group. However, when diagnostic technologies are used specifically for detection of activity of the HHV-6, a strong correlation between HHV-6 and the pathogenesis of MS is observed. Our group has recently investigated the level of similarity between the envelope protein of HERV-W and MOG. A comparison of the envelope MOG identified five IgG-like domain of MOG-like extending the idea of the HERV-W may be involved in the immunopathogenesis of MS, perhaps to facilitate recognition by the immune system MOG retroviral regions. We have also shown that most patients showed expression of the HERV-W envelope at some level. Nine of the ten tested samples had medium to high levels of HERV-W envelope expression against very low expression levels or no activity in healthy controls, confirming the association between MS activity and HERV-W in our population.

A recent study in Italy showed that EBV stimulates the expression of HERV-W in cells from blood and brain in vitro. They suggest that the pathogenesis of MS, a possible model could include EBV as the initial trigger of MS, years later, and shows the HERV-W as real to pathogenicity of MS, in striking parallel with the behavior of the disease in their remitting form contributor the appellant.

Objectives:

Primary Objective: correlate clinical and imaging of MS activity with quantitative assessment of HERV-W and viruses of the Herpesviridae family in the blood of patients with MS.

Secondary Objective:

Assess expression of HERV-W and Herpesvirus and compare the viruses expression among patients with MS and healthy controls with and without other neurological diseases.

Significance:

MS is a multifactorial disease, with genetic and environmental etiology. It is great the interest the researchers in associated factors to establish a causal relationship. Several viruses have been linked to the pathogenesis and disease activity. Although herpesvirus and HERV-W viruses are the most important in the attempt to establish a causal relationship and with activity of MS, until now there are many questions that remain open about the role of these viruses in the etiology and development of disease.

Hypothesis:

With this work it is expected to find more possible answers on the etiopathogenesis and inflammatory activity related to MS, and thus, provide more consistent data that will help the formulation of increasingly specific and effective therapies directed to this pathology.

Methods:

Initially, all samples will be analyzed by ELISA immunoassay for the detection of IgG and immunoglobulin M (IgM) anti-EBV and CMV antibodies in the serum of the participants, using commercial kits.

The nucleic acid extraction will be performed (DNA and RNA), according to manufacturer's instructions. All protocols to ensure the purity of the RNA and absence of DNA in the samples will be adopted in the analyze of expression (and thus detection of transcripts). Thus, the nucleic acids are subjected to treatment with DNAse and verification by RT-PCR HERV-W. Only samples containing RNA will be transcribed and subjected to further analysis. RNA quantification of the HERV-W will be made on mononuclear cells (PBMC) by a quantitative polymerase chain reaction (qRT-PCR) specific for the subtype MSRV of the HERV-W family.

The detection of herpesvirus DNA will initially be made by a PCR, using two sets of primers (HSVPAN and VZVPAN). After amplification is carried out an enzymatic digestion with BamHI and BstUI for typing the herpesvirus eight types including human herpesvirus 6 (6A and 6B). For samples that prove positive, a qRT-PCR will be held for specific viruses.

Design:

A prospective, longitudinal study that collected biological material and the presence of a control group will be held. This project will be analyzed by the individuals, through the term of free and informed consent. Only by signing the consent form the patient will be able to participate in this survey.

Blood samples of patients from the neurology outpatient clinic (CATEM and other specialties) will be done during routine visit by a qualified professional. The blood of the patients from the Blood Bank will be collected in conjunction with the examination routinely performed. All materials collected will be sent to the virology laboratory at the Institute of Tropical Medicine, University of São Paulo, where laboratory tests are performed.

Patients will be assessed for degree of clinical and imaging disease activity by analyzing annualized rate of relapses, EDSS-scale increases and increased cranial lesions on MRI and disease activity classified as MILD, MODERATE and SEVERE according to the proposed criteria by Freedman et al. The cranial MRI will be performed only for groups with MS and with other neurological diseases.

Statistical Methods:

After laboratory test results, data will be analyzed and receive necessary treatment for its statistical interpretation and comparison with the activity of disease using parametric and non-parametric tools. The Student-t and Mann-Whitney tests will be used to evaluate associations between clinical, demographic and laboratory parameters. The significance level of alpha = 0.05 or 5% to reject the null hypothesis will be fixed.

Sample Size Calculation:

The sample size was determined based on the percentage of the population with and without MS showing detectable expression of HERV-W in PBMC. Although the number of patients with MS that exhibits activity retrovirus envelope is close to 95%, we assume more conservative values for the sample calculation. Therefore, assuming expression by 50% and 10% for cases and controls, respectively, a sample size of 28 cases and 28 controls is necessary, based on a confidence level = 95% power to detect 80%, according to the Kelsey-method. Thus, as the investigators will analyze three groups (with MS, without MS and other neurological diseases) the total N is 84 subjects, 28 per group.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with multiple sclerosis;
* patients diagnosed with other neurological diseases (Lateral Amniotrofic Sclerosis , Headache, Parkinson's, Dementia and Epilepsy);
* healthy control: blood donors;

Exclusion Criteria:

* patients diagnosed with other non-neurological diseases;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study group will be composed by patients diagnosed with multiple sclerosis and with other neurological diseases ( Lateral AmniotroficSclerosis, Headache, Parkinson's, Dementia and Epilepsy). And the control group will be composed by blood donors who are considered healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Composite: Degree of disease activity | 1 year
  The degree of disease activity will be a composite of clinical and imaging measures. Clinical measures will be analyzed by annualized rate of relapses and EDSS-scale increase. The imaging measures will be analyzed by increase cranial lesions on MRI. This date will be correlated with quantitative assessment of HERV-W and viruses of the Herpesviridae family.

REFERENCES:
- [Result] Lassmann H, Bruck W, Lucchinetti C. Heterogeneity of multiple sclerosis pathogenesis: implications for diagnosis and therapy. Trends Mol Med. 2001 Mar;7(3):115-21. doi: 10.1016/s1471-4914(00)01909-2. PMID 11286782
- [Result] Martin R, McFarland HF. Immunological aspects of experimental allergic encephalomyelitis and multiple sclerosis. Crit Rev Clin Lab Sci. 1995;32(2):121-82. doi: 10.3109/10408369509084683. PMID 7598789
- [Result] Steinman L. Multiple sclerosis: a coordinated immunological attack against myelin in the central nervous system. Cell. 1996 May 3;85(3):299-302. doi: 10.1016/s0092-8674(00)81107-1. No abstract available. PMID 8616884
- [Result] Sun JB, Olsson T, Wang WZ, Xiao BG, Kostulas V, Fredrikson S, Ekre HP, Link H. Autoreactive T and B cells responding to myelin proteolipid protein in multiple sclerosis and controls. Eur J Immunol. 1991 Jun;21(6):1461-8. doi: 10.1002/eji.1830210620. PMID 1710567
- [Result] Bernard CC, de Rosbo NK. Immunopathological recognition of autoantigens in multiple sclerosis. Acta Neurol (Napoli). 1991 Apr;13(2):171-8. PMID 1891982
- [Result] Sellebjerg F, Christiansen M, Garred P. MBP, anti-MBP and anti-PLP antibodies, and intrathecal complement activation in multiple sclerosis. Mult Scler. 1998 Jun;4(3):127-31. doi: 10.1177/135245859800400307. PMID 9762660
- [Result] Egg R, Reindl M, Deisenhammer F, Linington C, Berger T. Anti-MOG and anti-MBP antibody subclasses in multiple sclerosis. Mult Scler. 2001 Oct;7(5):285-9. doi: 10.1177/135245850100700503. PMID 11724443
- [Result] Hellings N, Baree M, Verhoeven C, D'hooghe MB, Medaer R, Bernard CC, Raus J, Stinissen P. T-cell reactivity to multiple myelin antigens in multiple sclerosis patients and healthy controls. J Neurosci Res. 2001 Feb 1;63(3):290-302. doi: 10.1002/1097-4547(20010201)63:33.0.CO;2-4. PMID 11170179
- [Result] Genain CP, Cannella B, Hauser SL, Raine CS. Identification of autoantibodies associated with myelin damage in multiple sclerosis. Nat Med. 1999 Feb;5(2):170-5. doi: 10.1038/5532. PMID 9930864
- [Result] Bernard CC, Johns TG, Slavin A, Ichikawa M, Ewing C, Liu J, Bettadapura J. Myelin oligodendrocyte glycoprotein: a novel candidate autoantigen in multiple sclerosis. J Mol Med (Berl). 1997 Feb;75(2):77-88. doi: 10.1007/s001090050092. PMID 9083925
- [Result] Genain CP, Hauser SL. Creation of a model for multiple sclerosis in Callithrix jacchus marmosets. J Mol Med (Berl). 1997 Mar;75(3):187-97. doi: 10.1007/s001090050103. PMID 9106075
- [Result] 't Hart BA, van Meurs M, Brok HP, Massacesi L, Bauer J, Boon L, Bontrop RE, Laman JD. A new primate model for multiple sclerosis in the common marmoset. Immunol Today. 2000 Jun;21(6):290-7. doi: 10.1016/s0167-5699(00)01627-3. PMID 10825741
- [Result] Owens GP, Gilden D, Burgoon MP, Yu X, Bennett JL. Viruses and multiple sclerosis. Neuroscientist. 2011 Dec;17(6):659-76. doi: 10.1177/1073858411386615. PMID 22130640
- [Result] Blond JL, Beseme F, Duret L, Bouton O, Bedin F, Perron H, Mandrand B, Mallet F. Molecular characterization and placental expression of HERV-W, a new human endogenous retrovirus family. J Virol. 1999 Feb;73(2):1175-85. doi: 10.1128/JVI.73.2.1175-1185.1999. PMID 9882319
- [Result] Komurian-Pradel F, Paranhos-Baccala G, Bedin F, Ounanian-Paraz A, Sodoyer M, Ott C, Rajoharison A, Garcia E, Mallet F, Mandrand B, Perron H. Molecular cloning and characterization of MSRV-related sequences associated with retrovirus-like particles. Virology. 1999 Jul 20;260(1):1-9. doi: 10.1006/viro.1999.9792. PMID 10405350
- [Result] Dolei A, Serra C, Mameli G, Pugliatti M, Sechi G, Cirotto MC, Rosati G, Sotgiu S. Multiple sclerosis-associated retrovirus (MSRV) in Sardinian MS patients. Neurology. 2002 Feb 12;58(3):471-3. doi: 10.1212/wnl.58.3.471. PMID 11839854
- [Result] Serra C, Sotgiu S, Mameli G, Pugliatti M, Rosati G, Dolei A. Multiple sclerosis and multiple sclerosis-associated retrovirus in Sardinia. Neurol Sci. 2001 Apr;22(2):171-3. doi: 10.1007/s100720170019. PMID 11603622
- [Result] Sotgiu S, Serra C, Mameli G, Pugliatti M, Rosati G, Arru G, Dolei A. Multiple sclerosis-associated retrovirus and MS prognosis: an observational study. Neurology. 2002 Oct 8;59(7):1071-3. doi: 10.1212/wnl.59.7.1071. PMID 12370465
- [Result] Perron H, Gratacap B, Lalande B, Genoulaz O, Laurent A, Geny C, Mallaret M, Innocenti P, Schuller E, Stoebner P, et al. In vitro transmission and antigenicity of a retrovirus isolated from a multiple sclerosis patient. Res Virol. 1992 Sep-Oct;143(5):337-50. doi: 10.1016/s0923-2516(06)80122-6. PMID 1282730
- [Result] Perron H, Firouzi R, Tuke P, Garson JA, Michel M, Beseme F, Bedin F, Mallet F, Marcel E, Seigneurin JM, Mandrand B. Cell cultures and associated retroviruses in multiple sclerosis. Collaborative Research Group on MS. Acta Neurol Scand Suppl. 1997;169:22-31. doi: 10.1111/j.1600-0404.1997.tb08146.x. PMID 9174637
- [Result] Christensen T, Tonjes RR, zur Megede J, Boller K, Moller-Larsen A. Reverse transcriptase activity and particle production in B lymphoblastoid cell lines established from lymphocytes of patients with multiple sclerosis. AIDS Res Hum Retroviruses. 1999 Feb 10;15(3):285-91. doi: 10.1089/088922299311466. PMID 10052759
- [Result] Garson JA, Tuke PW, Giraud P, Paranhos-Baccala G, Perron H. Detection of virion-associated MSRV-RNA in serum of patients with multiple sclerosis. Lancet. 1998 Jan 3;351(9095):33. doi: 10.1016/s0140-6736(98)24001-3. No abstract available. PMID 9433428
- [Result] Sotgiu S, Arru G, Mameli G, Serra C, Pugliatti M, Rosati G, Dolei A. Multiple sclerosis-associated retrovirus in early multiple sclerosis: a six-year follow-up of a Sardinian cohort. Mult Scler. 2006 Dec;12(6):698-703. doi: 10.1177/1352458506070773. PMID 17262996
- [Result] Sotgiu S, Mameli G, Serra C, Zarbo IR, Arru G, Dolei A. Multiple sclerosis-associated retrovirus and progressive disability of multiple sclerosis. Mult Scler. 2010 Oct;16(10):1248-51. doi: 10.1177/1352458510376956. Epub 2010 Aug 4. PMID 20685761
- [Result] Perron H, Mekaoui L, Bernard C, Veas F, Stefas I, Leboyer M. Endogenous retrovirus type W GAG and envelope protein antigenemia in serum of schizophrenic patients. Biol Psychiatry. 2008 Dec 15;64(12):1019-23. doi: 10.1016/j.biopsych.2008.06.028. Epub 2008 Aug 29. PMID 18760403
- [Result] Mameli G, Poddighe L, Astone V, Delogu G, Arru G, Sotgiu S, Serra C, Dolei A. Novel reliable real-time PCR for differential detection of MSRVenv and syncytin-1 in RNA and DNA from patients with multiple sclerosis. J Virol Methods. 2009 Oct;161(1):98-106. doi: 10.1016/j.jviromet.2009.05.024. Epub 2009 Jun 6. PMID 19505508